CLINICAL TRIAL: NCT06888843
Title: A Single-center, Open-label, Randomized Phase II Study to Evaluate the Use of Capecitabine in Monotherapy and in Combination With Oxaliplatin in Elderly Patients as Adjuvant Chemotherapy for Locally Advanced Colorectal Cancer.
Brief Title: Study to Evaluate the Use of Capecitabine in Monotherapy and in Combination With Oxaliplatin in Elderly Patients as Adjuvant Chemotherapy for Locally Advanced Colorectal Cancer.
Acronym: AHTCRR-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nizhny Novgorod Regional Clinical Oncology Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRR-2025
Record Dates: First submitted 2025-03-06; First posted 2025-03-21 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
Keywords: XELOX; Capecitabine; Overall survival; Disease free survival; Toxicity profile; Comprehensive geriatric evaluation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment All patients with locally advanced colorectal cancer after radical surgical intervention who have not previously received systemic antitumor treatment will be randomized into two groups receiving fluoropyrimidines in mono-regimen and in combination with oxaliplatin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoropyrimidines in mono-regimen (Experimental): Capecitabine 2000mg/m2 per day, orally from day 1 to 14, 1 week break. Cycle of 21 days (start the next course on day 22).
  Interventions: Drug: Capecitabine
- Combination chemotherapy based on platinum preparations (Experimental): XELOX: Oxaliplatin 100-130mg/m2 w/v #1 on day 1 + Capecitabine 2000mg/m2 per day, orally from day 1 to 14, 1 week break.
  Cycle of 21 days (start of the next course on day 22).
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 2000mg/m2 from day 1 to 14
Drug: Oxaliplatin — Oxaliplatin 130mg/m2 on day 1, cycle of 21 days
  Arms: Combination chemotherapy based on platinum preparations

SUMMARY:
All patients with locally advanced colorectal cancer after radical surgical intervention who have not previously received systemic antitumor treatment will be randomized into two groups receiving fluoropyrimidines in mono-regimen and in combination with oxaliplatin.

Main objectives:

* to compare the 3-year disease-free survival and 5-year overall survival rates in the two groups.
* to identify, through a comprehensive geriatric assessment among elderly patients, the groups that benefit most from adjuvant chemotherapy.

Patients will be treated until progression of the process is detected or the maximum effect of therapy is reached (the longest duration of treatment is 6 months).

DETAILED DESCRIPTION:
The study is a single-center, open-label, randomized Phase II study. The study will be divided into a screening phase (4 weeks prior to inclusion in the study), a treatment phase (up to 6 months) and a long-term follow-up phase (up to 28 days from the end of treatment - follow-up to assess the safety of therapy, up to 3 years from the end of treatment to assess survival and follow-up).

During the screening phase, patients with MR CRC will undergo examinations to fulfill the inclusion and exclusion criteria for the study.

Next, elderly patients meeting these criteria-who have locally advanced colorectal cancer-will be randomized in a ratio of approximately 1:1 into 2 groups.

The study is planned to include 160 patients, 80 in each group, for a total of 160 patients.

Patient groups

1. Capecitabine in mono-regimen
2. PCT according to XELOX regimen Stratification factors - gender m/f, age <75 />75, presence of postoperative complications yes/no.

The patients will be treated until the progression is detected or the maximum effect of therapy is achieved (the longest duration of treatment is 8 cycles). At the end of the treatment period, all patients will enter the observation phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age 70 years and older;
2. Obtaining informed consent to participate in the study;
3. Morphologically confirmed diagnosis of colorectal cancer;
4. Stage III colorectal cancer;
5. Underwent radical surgical intervention for primary colorectal tumor;
6. ECOG score of 0 - I;
7. Life expectancy of more than 6 months;
8. No history of systemic drug therapy for CRC;
9. Adequate liver, kidney and bone marrow function;
10. Absence of severe uncontrolled concomitant chronic diseases and acute illnesses.

Exclusion Criteria:

1. Having previously received any systemic therapy for CRC;
2. Time after surgical treatment of more than 12 weeks;
3. Stage I-II and IV disease;
4. Confirmed dihydropyrimidine dehydrogenase deficiency in blood by PCR (alteration of alleles c.[190511G > A], c.[1679T >G],[2846A > T], [1129-5923C >G], [c.1236 G>A(HapB3)]);
5. Severe uncontrolled comorbid chronic diseases or acute illnesses;
6. Presence of a second malignancy (except for previously cured malignancies);
7. Any condition that, in the opinion of the physician, would interfere with the study procedures.

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
The disease free survival | 3 years
  Time from randomization to disease recurrence

SECONDARY OUTCOMES:
The overall survival | 5 years
  Time from randomization to death from any cause or date of last observation in the absence of these events. In months with an accuracy of 0.1.
Аssessment of the quality of life | 5 years
  Quality of life assessment by European Organisation for Research and Treatment of Cancer scale Quality of Life Questionnaire - Core 30 (QLQ-C30) by Scoring of the QLQ-C30 Summary Score using the descriptive analysis with the qlqc30 command (detailed description in manual ISBN 2-9300 64-22-6).
Toxicity assessment | 6 months
  Treatment toxicity according to common terminology criteria for adverse events version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Gamayunov, DMS, Study Director — Study Director
Locations (1):
- Research Institute of Clinical Oncology "Nizhny Novgorod Regional Clinical Oncological Dispensary", Nizhny Novgorod, Russia

IPD SHARING:
Plan to Share IPD: No